CLINICAL TRIAL: NCT03983564
Title: Derivation and Validation of a Combination of BOSTON Score and DES-OSA Score for Selection of OSA Patients. A Preliminary Study.
Brief Title: Derivation and Validation of a Combination of BOSTON Score and DES-OSA Score for Selection of OSA Patients.
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, Head of Department, Astes
Other Study IDs: PS-PSG
Record Dates: First submitted 2019-06-06; First posted 2019-06-12 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: Patients in this group will serve to validate the cutoff of the combination of the DES-OSA and BOSTON scores derived in the retrospective group.
  Interventions: Other: Cutoff Validation

INTERVENTIONS:
Other: Cutoff Validation — We will validate the cutoff of the combination of BOSTON score and DES-OSA scores with the result of a polysomnography.

SUMMARY:
Derivation and Validation of a combination of BOSTON score and DES-OSA score to exclude OSA or to confirm OSA in patients.

DETAILED DESCRIPTION:
The aim of this study is to derive and to validate a combination of BOSTON score and DES-OSA score.

Firstly, the investigators will use a retrospective cohort of 400 patients to determine this combination. It will allow classifying patients in 3 groups: 1) patients for whom OSA can be excluded with certitude, 2) patients for whom OSA can be diagnosed with certitude, and 3) an intermediate group.

Secondly, the 100 patients included in this study will serve to validate the cutoff of the abovementioned combination into a new population.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted in the Clinique Saint-Luc of Bouge for a polysomnography

Exclusion Criteria:

* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population to validate the cutoff of the combination of scores
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Validation of cutoff values for the combination of BOSTON score and DES-OSA score in order to classify patients following their risk to present an OSA Syndrome. | One month
  Validation of cutoff values for the combination of BOSTON score and DES-OSA score derived in the retrospective group in order to validate these cutoff values in order to classify patients following their risk to present an OSA (Obstructive Sleep Apnea) Syndrome. The measurements will serve to validate the classification establish in the retrospective study, namely 1) patients without OSA with certitude, 2) patients with OSA with certitude, 3) an intermediate category.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, MD, PhD, Principal Investigator — Clinique Saint-Luc of Bouge
Locations (1):
- Clinique Saint-Luc de Bouge, Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No
No sharing